CLINICAL TRIAL: NCT06622135
Title: Development of a Home Test for Measuring Plasma P-tau217 in Alzheimer's Disease Using Tasso Lancet Device
Brief Title: Home Test for Measuring Plasma P-tau217 in Alzheimer's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Insight Research Institute (Other)
Responsible Party: Principal Investigator, Abeer Gharaibeh, Director of Research, Insight Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU24080011
Record Dates: First submitted 2024-09-19; First posted 2024-10-01 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease; Healthy Subjects
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Blood draw using IV and at home device (Other)
  Interventions: Device: Tasso Lancet Device

INTERVENTIONS:
Device: Tasso Lancet Device — blood samples will be obtained from all participants using Tasso device

SUMMARY:
The goal of this is to develop an easy at home test that can be used to assist in diagnosing Alzheimer's disease (AD). The test will use an FDA approved device for at home blood sample collection. The blood samples will be evaluated to determine if the concentration of p-tau217, a biomarker that is elevated in AD patients, measured from blood samples collected using the at home device is comparable to the results obtained from blood samples collected by venipuncture.

ELIGIBILITY:
Inclusion Criteria:

* Subject with Alzheimer's Disease Only: diagnosed according the NIA-AA diagnostic AD criteria
* Healthy Control Only: Subject does not have history of cognitive impairment
* 55 - 90 years old
* Subject able to comply with study procedures
* Subjects must be able to use the Tasso device for blood sample collection as per the provided instructions (can be performed with the assistance of a caregiver)
* Subjects must be able to undergo IV sampling
* Have a study partner who will provide written informed consent to participate, and assist with blood collection when applicable

Exclusion Criteria:

* Subjects with systemic conditions which were not adequately controlled through a stable medication regimen
* Subjects with any known significant bleeding disorders or conditions that contraindicate blood sample collection (e.g., hemophilia, severe thrombocytopenia)
* Subjects with a known history of severe skin allergies or reactions to adhesives (since the Tasso device involves adhesive application to the skin)
* Subjects currently taking anticoagulant or antiplatelet medications that could interfere with blood collection or increase the risk of complications
* Subjects who have undergone major surgery or have been hospitalized for any reason in the last 3 months prior to study enrollment
* Participation in a clinical study within the 2 month

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2024-12-07 (Actual); Study Completion 2024-12-07 (Actual)

PRIMARY OUTCOMES:
Agreement between measurements of P-tau217 concentration in blood samples from Tasso device and venipuncture | Day 1

SECONDARY OUTCOMES:
Means of p-tau217 concentration in subjects with and without AD | Day 1
Agreement between measurements of P-tau217 concentration by the ALZpath P-tau217 and Janssen P-tau217+ assays | Day 1
Percentage of Tasso devices which are loss, damaged, or with inadequate blood volume for analysis | Day 1
Mean fold-change of p-tau217 concentration in subjects with and without AD | Day 1
Effect size of p-tau217 concentration in subjects with and without AD | Day 1

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Insight Research Institute/Insight Hospital and Medical Center Chicago, Chicago, Illinois
  - Insight Research Institute, Flint, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Deidentified Data will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code